CLINICAL TRIAL: NCT00579215
Title: Lung Cancer Informational Study (LCIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Virginia (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Leslie Tyson, NP, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-141
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Cancer; Enhanced Care; Decision-Making; Advance Lung Cancer; Stage III Lung Cancer; Stage IV Lung Cancer
Keywords: Cancer; Enhanced Care; Decision-Making; Advance Lung Cancer; Questionaires; Stage III Lung Cancer; Stage IV Lung Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

ARMS (2):
- 1 (Experimental): Enhance Care (EC) will receive a decision aid with seven components: social support, anticipatory guidance, adhering to the patient's preference for participation in treatment decision making, a quality decision-making process tutorial, normalization (using a CD program), structured time with oncology professionals to discuss difficult decisions, and values clarification of 3 decisions throughout treatment. Self-report measures will be used for all participants in addition to probes for the taped interviews with EC. The outcome measures are quality decision making and decisional conflict. Two panels (decision making and lung cancer) will review the protocol twice. The plan will include serially screening the appointment roster. The decision aid will be administered during three clinic visits.
  Interventions: Behavioral: Enhance Care
- 2 (Other): As an intentional control, the usual care group will receive standard care related to lung cancer and treatment; they will not receive any oral, written, or recorded information related to decision making. Usual care includes anticipatory guidance related to the disease and treatment (e.g., what to do about treatment side effects, signs of an infection, why a treatment would be changed or stopped) using patient education materials normally used in the MSKCC, TOS, Outpatient Clinic.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Enhance Care — EC will receive a decision aid with seven components: social support, anticipatory guidance, adhering to the patient's preference for participation in treatment decision making, a quality decision-making process tutorial, normalization (using a CD program), structured time with oncology professionals to discuss difficult decisions, and values clarification of 3 decisions throughout treatment. Self-report measures will be used for all participants in addition to probes for the taped interviews with EC. The outcome measures are quality decision making and decisional conflict. Two panels (decision making and lung cancer) will review the protocol twice. The plan will include serially screening the appointment roster. The decision aid will be administered during three clinic visits
  Other Names: EC
  Arms: 1
Behavioral: Usual Care — As an intentional control, the usual care group will receive standard care related to lung cancer and treatment; they will not receive any oral, written, or recorded information related to decision making. Usual care includes anticipatory guidance related to the disease and treatment (e.g., what to do about treatment side effects, signs of an infection, why a treatment would be changed or stopped) using patient education materials normally used in the MSKCC, TOS, Outpatient Clinic.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate a new program to help the patient and the caregiver make decisions about treatment for lung cancer. We need to know if a new information program is helpful to patients. The way that we will do this is by comparing it with the usual information program that we now provide.

Patient are asked to make difficult decisions about their treatments. These decisions may include when to change treatments or when to stop treatment altogether. Most patients ask a family member or close friend to help them with these difficult decisions. A "caregiver" is someone they can count on to give support (either emotional or physical) over a period of time. The doctors and nurses will also help patients and their caregiver to make these decisions.

They will tell them the risks with each treatment, the success with each treatment, and how much time there is for making each decision.

DETAILED DESCRIPTION:
Many patients with advanced lung cancer and their caregivers struggle with treatment decisions, such as when to say "enough." Patient preparation for facing termination of cancer-directed therapy for the number one cause of cancer mortality for both men and women in the U.S. is not well handled in most clinical practices. Sparse literature validates that this concern is often denied by investigators. Failure to engage in a systematic, informed decision-making process, even in the initial stage of treatment, may often result in patients looking back and saying, "Knowing what I know now, I wouldn't make the same choice" The long-term goal of this program of research is to enhance patient care for lung cancer by oncology health professionals and to promote patient empowerment to make informed choices, defined as the ability to actively understand and influence one's health status. For this study, shared decision making is defined as a tailored, interactive process (emphasizing beliefs/personal values) in which the patient is informed enough to ask pertinent questions and to participate in the final decision at his/her own preference and comfort levels. The intent is to test a decision aid for patients with advanced lung cancer to help facilitate informed decisions about treatments that affect quality of life, including termination of cancer-directed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically determined non-small cell lung cancer
* Stage IIIA, IIIB or IV extent
* No prior chemotherapy unless used in adjuvant therapy, completed more than two years ago, and no sign of any other malignancy active at this time
* Lung cancer-directed treatment with a standard or investigative chemotherapy regimen at entry
* Patients with brain metastasis are acceptable provided they are at least 3 weeks from completion of radiation therapy for brain metastasis, have stable and acceptable neurological status, and meet all other eligibility criteria. For patients undergoing gamma knife procedure, cognitive ability is the judgment call of the oncologist and study nurse as to whether comprehension is not a problem.

Exclusion Criteria:

* Performance status of KPS 60-100% or ECOG 0-2;
* No age limit
* Life expectancy greater than three months
* A caregiver (any family member or concerned other who consistently provides emotional and/or physical support) available to also participate
* Patient and caregiver are able to understand English (ability to repeat back in their own words)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of implementing a short, clinic-based, decision-making aid (cognitive-behavioral skills intervention) for patients with advanced lung cancer (and their caregivers) facing cancer-directed treatment. | 2 years

SECONDARY OUTCOMES:
To gather data for testing the hypothesis that patients with advanced lung cancer who receive a decision aid will report increased quality decision making, and decreased decisional conflict at the end of Decision 3 compared to the usual care group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leslie B Tyson, NO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Virginia- School of Nursing, Charlottesville, Virginia

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org